CLINICAL TRIAL: NCT03904836
Title: Pharmacokinetics of Tobramycin Administered at the Beginning of Intermittent Hemodialysis Session
Brief Title: Tobramycin Administered at the Beginning of Dialysis
Acronym: ESRD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Jean-Philippe Lafrance, Principal Investigator, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-1619
Record Dates: First submitted 2019-02-08; First posted 2019-04-05 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Renal Dialysis; Renal Failure, Chronic
Keywords: Chronic Renal Diseases; Kidney Failure, Chronic; Renal Failure, Chronic; Tobramycin; Aminoglycosides; Pharmacokinetics; Infection; Anti-Bacterial Agents; Antibiotics; Renal Insufficiency, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Infections | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tobramycin (Experimental): Subjects with end-stage renal disease who have been involved in an intermittent hemodialysis program and who have suspected or diagnosed Gram-negative rod-type infection
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Tobramycin — 5 milligrams per kilogram intravenous for one dose

SUMMARY:
The purpose of the study is to evaluate whether the administration of a full tobramycin dose (5 mg/kg) during the first 30 minutes of a hemodialysis session provides favorable pharmacokinetic parameters in subjects with end-stage renal disease who are suspected or has been diagnosed with Gram-negative rod-type infection.

It is anticipated that the administration of a single 5 mg/kg dose of tobramycin during the first 30 minutes of a hemodialysis session will achieve an optimal ratio of maximum tobramycin concentration to minimal inhibitory concentration (Cmax/CMI) of 8 to 10 while limiting the accumulation (trough < 2 mg/L before the next hemodialysis session) in end-stage renal disease subjects requiring intermittent hemodialysis sessions.

DETAILED DESCRIPTION:
STUDY DESIGN:

Prospective, monocentric, non-randomized, uncontrolled pharmacokinetic study

End-stage renal disease subjects who have been involved in an intermittent hemodialysis program and who have suspected or diagnosed Gram-negative rod-type infection.

Pharmacokinetic parameters: Tobramycin concentration analyses done at the beginning of hemodialysis session (before tobramycin administration), 30 minutes after completion of the infusion (will allow us to calculate the peak), during hemodialysis session (additional), at the end of hemodialysis session, between hemodialysis sessions (optional) and just before the next hemodialysis session (will allow us to analyse the trough).

RECRUITMENT PROCESS:

A systematic daily screening for hemodialysis hospitalized subjects or subjects followed at the outpatient clinic who have a suspicion or diagnosis of Gram-negative rod type infection will be made by the research coordinators. Software routinely used in the clinic at Maisonneuve-Rosemont Hospital (Gesphar, NumeRx, Oacis and Medurge) will be used to ensure the identification of potential subjects. The pharmacists responsible for validation of prescriptions at the pharmacy department will collaborate with the research team to help identifying eligible candidates. An eligibility assessment tool will be used and subjects who meet the inclusion criteria and do not meet any exclusion criteria will be considered as eligible candidates. Thereafter, additional baseline information will be collected from the medical file (e.g. ethnicity) or by questioning the subject. A member of the research team will addressed the eligible subject, will explain the study and present the Information Form and Informed Consent (FIC), that will document informed consent of the subject.

DATA COLLECTION:

A minimum of four blood samples and a maximum of six blood samples will be collected. The sampling scheme is as follows: at the beginning of hemodialysis session (before tobramycin administration), 30 minutes after completion of the infusion, during hemodialysis session (additional), at the end of hemodialysis session, between hemodialysis sessions (optional) and just before the next hemodialysis session.

A member of the research team will provide the tubes to the nursing, will write sampling times and will ship the blood samples to the laboratory.

STUDY SAMPLE:

Since the objective is to obtain robust pharmacokinetic parameters, the calculation of the sample size aims at a sufficient number of participants to obtain a convergence of facilitated pharmacokinetic parameters, thus obtaining values of coefficients of variation of less than 40%, while maintaining a statistical power of 80%. The calculation uses the variability of the parameters obtained by Veinstein et al. In this study, the residual clearance (Clnhd) is the parameter with the greatest variability (average of 10.4 mL / min with a standard deviation of 6.4 mL / min). Thus, the variability used in calculating the sample size is that of the parameter with the greatest variability, the residual clearance. The sample studied by Veinstein et al. not having the same characteristics as the subjects of the study, the variability could be greater than the reference sample and a safety margin of 30% is added. A total of 12 subjects to be recruited is therefore planned. No correction is applied for losses at the follow-up or withdrawal of consent considering the short duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 and over;
* Subjects with end-stage renal disease who are on an intermittent hemodialysis program (three times a week, 3-4 hours) at the Hôpital Maisonneuve-Rosemont hemodialysis unit for at least one month;
* Subjects with suspicion or diagnosis of Gram-negative rod-type bacteria infection for which an antibiotic is prescribed;
* Subjects able to consent to the study (consent form read and signed by the subject).

Exclusion Criteria:

* Contraindication or possible medical hazard related to the administration of tobramycin or to any ingredient in the formulation (e.g. sulphites), such as severe allergies or aminoglycoside-reported previous intolerances;
* Variable residual renal function (e.g. acute or transient renal failure requiring occasional hemodialysis sessions, post-renal transplantation);
* Conditions sensitive to the side effects of tobramycin (e.g. history of myasthenia gravis, Parkinson's disease, vestibular or auditory disorder);
* Subjects with impaired volume of distribution (ie, severe burns [> 20%], significant ascites, decompensation for acute heart failure requiring hospitalization, admission to the critical care unit, cystic fibrosis, morbid obesity [dry weight greater than 50% of ideal weight]);
* Pregnant or breastfeeding women;
* Unstable hemodynamic status (risk of not tolerating / completing a 3-4 hour dialysis session);
* Recent treatment with an aminoglycoside (<1 month);
* Participation in another research protocol;
* Inability to give free and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Ratio of maximum tobramycin concentration to minimal inhibitory concentration | The timeframe for data collection for this outcome is 48 hours to 72 hours
  In subjects receiving a single 5 mg/kg tobramycin dose during the first 30 minutes of a hemodialysis session, to determine the proportion of subjects in whom the maximum concentration is greater than or equal to 8 times that of the minimal inhibitory concentration

SECONDARY OUTCOMES:
Tobramycin trough level | The timeframe for data collection for this outcome is 48 hours to 72 hours
  In subjects receiving a single 5 mg/kg tobramycin dose during the first 30 minutes of a hemodialysis session, to determine the proportion of subjects whose trough concentration of tobramycin is less than or equal to 2 mg / L.
Residual clearance | The timeframe for data collection for this outcome is 48 hours to 72 hours
Clearance associated with hemodialysis | The timeframe for data collection for this outcome is 48 hours to 72 hours
Volume of distribution | The timeframe for data collection for this outcome is 48 hours to 72 hours
Total area under the curve | The timeframe for data collection for this outcome is 0 to 48 or 72 hours (depending on time between the two dialysis)
Area under the curve between 0 to 24h after administration | The timeframe for data collection for this outcome is 0 to 24 hours
Tobramycin concentration | The timeframe for data collection for this outcome is 24 hours to 72 hours
  Tobramycin concentration 24h, 48h and 72h after administration

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lafrance, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cheikh Hassan HI, Tang M, Djurdjev O, Langsford D, Sood MM, Levin A. Infection in advanced chronic kidney disease leads to increased risk of cardiovascular events, end-stage kidney disease and mortality. Kidney Int. 2016 Oct;90(4):897-904. doi: 10.1016/j.kint.2016.07.013. Epub 2016 Aug 31. PMID 27591084
- [Background] Kato S, Chmielewski M, Honda H, Pecoits-Filho R, Matsuo S, Yuzawa Y, Tranaeus A, Stenvinkel P, Lindholm B. Aspects of immune dysfunction in end-stage renal disease. Clin J Am Soc Nephrol. 2008 Sep;3(5):1526-33. doi: 10.2215/CJN.00950208. Epub 2008 Aug 13. PMID 18701615
- [Background] Reynvoet E, Vandijck DM, Blot SI, Dhondt AW, De Waele JJ, Claus S, Buyle FM, Vanholder RC, Hoste EA. Epidemiology of infection in critically ill patients with acute renal failure. Crit Care Med. 2009 Jul;37(7):2203-9. doi: 10.1097/CCM.0b013e3181a03961. PMID 19487937
- [Background] Eschenauer GA, Lam SW, Mueller BA. Dose Timing of Aminoglycosides in Hemodialysis Patients: A Pharmacology View. Semin Dial. 2016 May;29(3):204-13. doi: 10.1111/sdi.12458. Epub 2016 Jan 12. PMID 26756428
- [Background] Sandoz Canada Inc. Product monograph: Tobramycin injection USP. Boucherville, QC: Sandoz Canada Inc.; 2017.
- [Background] O'Shea S, Duffull S, Johnson DW. Aminoglycosides in hemodialysis patients: is the current practice of post dialysis dosing appropriate? Semin Dial. 2009 May-Jun;22(3):225-30. doi: 10.1111/j.1525-139X.2008.00554.x. Epub 2009 Apr 5. PMID 19386073
- [Background] ANSM. Bon usage des aminosides administrés par voie injectable: gentamicine, tobramycine, netilmicine, amikacine - Mise au point. Paris: National Security Agency of Medicines and Health Products; 2011.
- [Background] Lacy MK, Nicolau DP, Nightingale CH, Quintiliani R. The pharmacodynamics of aminoglycosides. Clin Infect Dis. 1998 Jul;27(1):23-7. doi: 10.1086/514620. PMID 9675444
- [Background] Moore RD, Lietman PS, Smith CR. Clinical response to aminoglycoside therapy: importance of the ratio of peak concentration to minimal inhibitory concentration. J Infect Dis. 1987 Jan;155(1):93-9. doi: 10.1093/infdis/155.1.93. PMID 3540140
- [Background] Brummett RE, Morrison RB. The incidence of aminoglycoside antibiotic-induced hearing loss. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):406-10. doi: 10.1001/archotol.1990.01870040028008. PMID 2317321
- [Background] Forge A, Schacht J. Aminoglycoside antibiotics. Audiol Neurootol. 2000 Jan-Feb;5(1):3-22. doi: 10.1159/000013861. PMID 10686428
- [Background] Gailiunas P Jr, Dominguez-Moreno M, Lazarus M, Lowrie EG, Gottlieb MN, Merrill JP. Vestibular toxicity of gentamicin. Incidence in patients receiving long-term hemodialysis therapy. Arch Intern Med. 1978 Nov;138(11):1621-4. doi: 10.1001/archinte.138.11.1621. PMID 309753
- [Background] Halmagyi GM, Fattore CM, Curthoys IS, Wade S. Gentamicin vestibulotoxicity. Otolaryngol Head Neck Surg. 1994 Nov;111(5):571-4. doi: 10.1177/019459989411100506. PMID 7970794
- [Background] Ahmed RM, Hannigan IP, MacDougall HG, Chan RC, Halmagyi GM. Gentamicin ototoxicity: a 23-year selected case series of 103 patients. Med J Aust. 2012 Jun 18;196(11):701-4. doi: 10.5694/mja11.10850. PMID 22554194
- [Background] Heintz BH, Thompson GR 3rd, Dager WE. Clinical experience with aminoglycosides in dialysis-dependent patients: risk factors for mortality and reassessment of current dosing practices. Ann Pharmacother. 2011 Nov;45(11):1338-45. doi: 10.1345/aph.1Q403. Epub 2011 Oct 18. PMID 22010003
- [Background] Dager WE, King JH. Aminoglycosides in intermittent hemodialysis: pharmacokinetics with individual dosing. Ann Pharmacother. 2006 Jan;40(1):9-14. doi: 10.1345/aph.1G064. Epub 2005 Dec 6. PMID 16332944
- [Background] Kamel Mohamed OH, Wahba IM, Watnick S, Earle SB, Bennett WM, Ayres JW, Munar MY. Administration of tobramycin in the beginning of the hemodialysis session: a novel intradialytic dosing regimen. Clin J Am Soc Nephrol. 2007 Jul;2(4):694-9. doi: 10.2215/CJN.01600407. Epub 2007 Jun 6. PMID 17699484
- [Background] Teigen MM, Duffull S, Dang L, Johnson DW. Dosing of gentamicin in patients with end-stage renal disease receiving hemodialysis. J Clin Pharmacol. 2006 Nov;46(11):1259-67. doi: 10.1177/0091270006292987. PMID 17050791
- [Background] Sowinski KM, Magner SJ, Lucksiri A, Scott MK, Hamburger RJ, Mueller BA. Influence of hemodialysis on gentamicin pharmacokinetics, removal during hemodialysis, and recommended dosing. Clin J Am Soc Nephrol. 2008 Mar;3(2):355-61. doi: 10.2215/CJN.02920707. Epub 2008 Jan 30. PMID 18235142
- [Background] Veinstein A, Venisse N, Badin J, Pinsard M, Robert R, Dupuis A. Gentamicin in hemodialyzed critical care patients: early dialysis after administration of a high dose should be considered. Antimicrob Agents Chemother. 2013 Feb;57(2):977-82. doi: 10.1128/AAC.01762-12. Epub 2012 Dec 10. PMID 23229487
- [Background] Venisse N, Dupuis A, Badin J, Robert R, Pinsard M, Veinstein A. Efficacy and safety of high-dose gentamicin re-dosing in ICU patients receiving haemodialysis. J Antimicrob Chemother. 2015 Jan;70(1):308-10. doi: 10.1093/jac/dku369. Epub 2014 Sep 19. No abstract available. PMID 25239463
- [Background] Dahlgren JG, Anderson ET, Hewitt WL. Gentamicin blood levels: a guide to nephrotoxicity. Antimicrob Agents Chemother. 1975 Jul;8(1):58-62. doi: 10.1128/AAC.8.1.58. PMID 1164007
- [Background] Lewis AS, Taylor G, Williams HO, Lewis MH. Comparison of venous and capillary blood sampling for the clinical determination of tobramycin serum concentrations. Br J Clin Pharmacol. 1985 Dec;20(6):597-601. doi: 10.1111/j.1365-2125.1985.tb05117.x. PMID 4091991
- [Background] Health Canada. Reporting Adverse Reactions to Marketed Health Products - Guidance Document for Industry. Health Canada; 2018
- [Background] Ariano RE, Zelenitsky SA, Kassum DA. Aminoglycoside-induced vestibular injury: maintaining a sense of balance. Ann Pharmacother. 2008 Sep;42(9):1282-9. doi: 10.1345/aph.1L001. Epub 2008 Jul 22. PMID 18648019
- [Background] Ding D, Liu H, Qi W, Jiang H, Li Y, Wu X, Sun H, Gross K, Salvi R. Ototoxic effects and mechanisms of loop diuretics. J Otol. 2016 Dec;11(4):145-156. doi: 10.1016/j.joto.2016.10.001. Epub 2016 Oct 27. PMID 29937824
- [Background] Jiang M, Karasawa T, Steyger PS. Aminoglycoside-Induced Cochleotoxicity: A Review. Front Cell Neurosci. 2017 Oct 9;11:308. doi: 10.3389/fncel.2017.00308. eCollection 2017. PMID 29062271
- [Background] Montreal east island integrated university health and social services center. Standard operating procedure: Tobramycin. Montreal: Maisonneuve-Rosemont Hospital; 2016.
- [Background] Boucher HW, Talbot GH, Bradley JS, Edwards JE, Gilbert D, Rice LB, Scheld M, Spellberg B, Bartlett J. Bad bugs, no drugs: no ESKAPE! An update from the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jan 1;48(1):1-12. doi: 10.1086/595011. PMID 19035777